CLINICAL TRIAL: NCT05511311
Title: Development of Frailty Prevention Clinic in Geriatric Comprehensive Clinic RSCM: The Role of Resistance Training as Sarcopenia and Frailty Management Towards Frailty Score, Sarcopenia Score, and Quality of Life
Brief Title: Development of Frailty Prevention Clinic in Geriatric Comprehensive Clinic RSCM:
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Siti Setiati, Prof, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Frailty Clinic
Record Dates: First submitted 2022-08-17; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Frailty; Sarcopenia; Resistance Training
Keywords: frailty; sarcopenia; elderly; resistance training
MeSH Terms: conditions — Frailty; Sarcopenia | interventions — Resistance Training; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): 12-week of Standard Therapy using elastic-band
  Interventions: Procedure: Standard Therapy
- Intervention (Experimental): 12-week of Resistance Training developed by RSCM using sand-bag
  Interventions: Procedure: Resistance Training

INTERVENTIONS:
Procedure: Resistance Training — Resistance training developed by the researcher (SCR-RSCM) for 12 weeks
  Arms: Intervention
Procedure: Standard Therapy — Standard therapy for 12 weeks
  Arms: Control

SUMMARY:
There is an increasing number of elderly population, not only in Indonesia, but also in the world. With increasing of age, there is also an increasing number of elderly with sarcopenia and frailty. Both of the diseases can lead to dependency, decrease quality of life, and morbidity. Besides nutrition, physical activity, especially resistance training is proven to be beneficial in improving sarcopenia and frailty condition.

Currently in Cipto Mangunkusumo National Hospital (RSCM), there is no comprehensive frailty prevention clinic in the geriatric inpatient clinics. This research can be the base of frailty and sarcopenia treatment in RSCM.

ELIGIBILITY:
Inclusion Criteria:

* Patients 60 years old or orlder
* Categorized as Pre-frail or Frail based on FRAIL criteria
* Is not in routine physical activity in the past 3 months
* Succeeded Mini Physical Performance Test with score 11 or more

Exclusion Criteria:

* Cognitive Disturbance (Abbreviated Mental Test < 8)
* Not consenting to join the trial

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Frailty Status | 12 weeks
  The FRAIL scale includes 5 components: Fatigue, Resistance, Ambulation, Illness, and Loss of weight (10). Frail scale scores range from 0-5 (i.e., 1 point for each component; 0=best to 5=worst) and represent frail (3-5), pre-frail (1-2), and robust (0) health status
Sarcopenia Status | 12 weeks
  Measured using:
  * BIA: <7.0 kg/m2 in men and <5.7 kg/m2 in women
  * Five times sit to stand: ≥12 seconds
  * Hand-grip strength: <28 kg for men and <18 kg for women
Walking Speed | 12 weeks
  <1.0 m/s
Patient's Quality of Life | 12 weeks
  Measured by EQ-5D: ranging from 0 ('worst imaginable health') to 100 ('best imaginable health')

SECONDARY OUTCOMES:
Prevalence of Frailty | 12 weeks
  The FRAIL scale includes 5 components: Fatigue, Resistance, Ambulation, Illness, and Loss of weight (10). Frail scale scores range from 0-5 (i.e., 1 point for each component; 0=best to 5=worst) and represent frail (3-5), pre-frail (1-2), and robust (0) health status
Prevalence of Sarcopenia | 12 weeks
  Measured using:
  * BIA: <7.0 kg/m2 in men and <5.7 kg/m2 in women
  * Five times sit to stand: ≥12 seconds
  * Hand-grip strength: <28 kg for men and <18 kg for women

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo National Hospital, Jakarta, Jakarta Pusat, Indonesia

REFERENCES:
- [Result] Chen LK, Woo J, Assantachai P, Auyeung TW, Chou MY, Iijima K, Jang HC, Kang L, Kim M, Kim S, Kojima T, Kuzuya M, Lee JSW, Lee SY, Lee WJ, Lee Y, Liang CK, Lim JY, Lim WS, Peng LN, Sugimoto K, Tanaka T, Won CW, Yamada M, Zhang T, Akishita M, Arai H. Asian Working Group for Sarcopenia: 2019 Consensus Update on Sarcopenia Diagnosis and Treatment. J Am Med Dir Assoc. 2020 Mar;21(3):300-307.e2. doi: 10.1016/j.jamda.2019.12.012. Epub 2020 Feb 4. PMID 32033882
- [Result] Mienche M, Setiati S, Setyohadi B, Kurniawan J, Laksmi PW, Ariane A, Tirtarahardja G. Diagnostic Performance of Calf Circumference, Thigh Circumference, and SARC-F Questionnaire to Identify Sarcopenia in Elderly Compared to Asian Working Group for Sarcopenia's Diagnostic Standard. Acta Med Indones. 2019 Apr;51(2):117-127. PMID 31383826
- [Result] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372